CLINICAL TRIAL: NCT01989364
Title: Multicenter Validation of Repetitive Functional Imaging in Locally Advanced Cervical Cancer
Brief Title: Repetitive Functional Imaging in Locally Advanced Cervical Cancer
Acronym: IMAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: The Netherlands Cancer Institute (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Jesper Kallehauge, Ph. D., Aarhus University Hospital
Other Study IDs: M-20100251
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background: The Apparent Diffusion Coefficient (ADC) acquired by Diffusion Weighted Imaging (DWI-MR) has been shown to correlate with cellular density. The ADC is indicative of Gross Tumour Volume (GTV), and preliminary data shows that the dynamics of DWI volumes during treatment (shrinkage) as well as dose to DWI volumes has impact on treatment outcome.

Hypoxic tumour cells within the primary tumour have been identified to have prognostic importance for local control Tumour hypoxia is caused by insufficiency of the tumour vasculature leading to both chronic diffusion limited and acute flow limited hypoxia. Radioresistant hypoxic cells diminish the rate of local control, and the hypoxia driven increase in metastatic potential of the tumour and lowers the rate of distant disease control. Functional imaging has the potential to visualise radioresistant tumour subvolumes. PET scanning (18F-FAZA) is hypothesized to visualise hypoxic tumour subvolumes, and dynamic contrast enhanced (DCE) MR imaging has been used to quantify the extent of poor perfusion regions within cervical tumours.

Objectives:

Primary:

Sensitivity and specificity of functional imaging (18F-FAZA PET (optional), T1w, T2w, DWI-MRI and DCE-MRI) to identify tumours with good and bad response to radio-chemotherapy

Secondary:

Determining whether there are differences in bias between centre. The difference in bias will be assessed for the T1 and T2 scans and the Ktrans and ADC maps.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced cervical cancer FIGO stage IB2-IV referred for definitive radio-chemotherapy.
* Patients where MR guided brachytherapy is part of standard patient treatment.
* Patients without previous record of allergic reaction to infusion of protocol related contrast media and tracers (Gadolinium-based for MR-imaging, FAZA (when performed))
* Patients with sufficient kidney function according to local regulations
* Patients of 18 years age and over.
* Cancer of the uterine cervix considered suitable for curative treatment.
* Positive biopsy showing Squamous cell carcinoma, Adeno cell carcinoma, Adeno Squamous cell carcinoma.
* Staging according to FIGO and TNM performed
* MRI pelvis at diagnosis available
* MRI, CT or PET-CT retroperitoneum and abdomen at diagnosis available
* MRI pelvis with applicator at Brachytherapy timepoint will be performed
* Patient informed consent

Exclusion Criteria:

* Patients with contra indications to MRI and FAZA-PET (when performed)
* Patients with active infection or severe medical condition
* Patients pregnant, lactating or with childbearing potential without adequate contraception.
* Other primary malignancies
* Metastatic disease beyond paraaortic region (L1-L2)
* Previous pelvic radiotherapy
* Previous total or partial hysterectomy
* Combination of preoperative radiotherapy with surgery
* Patients receiving Brachytherapy only
* Patients receiving External Beam radio therapy only
* Patients receiving neoadjuvant chemotherapy, hyperthermia or other antineoplastic treatments not approved by the Embrace study committee
* Contra indications to BT

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced cervical cancer eligible for chemo-radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-02 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Tumor volume | pre-treatment, week2, week5, week6, week 7

CONTACTS AND LOCATIONS:
Locations (3):
- University Hospitals Leuven, Leuven, Belgium
- Aarhus University Hospital, Aarhus, Denmark
- The Netherlands Cancer Institute, Amsterdam, Netherlands